CLINICAL TRIAL: NCT07270796
Title: A Phase I, Open-label, Randomized, Active-Controlled Trial to Evaluate the Safety and Immunogenicity of the DuoChol Oral Cholera Vaccine in 18 to 45 Years Old Healthy Participants in Sweden
Brief Title: Safety and Immunogenicity Study of the DuoChol Oral Cholera Vaccine in Healthy Participants
Acronym: DuoChol
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: International Vaccine Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IVI DuoChol 001; 226726/Z/22/Z (Other Grant/Funding Number: Wellcome Trust); 2025-522633-57-00 (EU CTIS Number)
Record Dates: First submitted 2025-11-18; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Cholera Vaccination Reaction
Keywords: Oral Cholera Vaccine; DuoChol; Phase 1 Trial; V. cholerae O1 Inaba; V. cholerae O1 Ogawa; recombinant cholera toxin B-subunit
MeSH Terms: interventions — Dukoral

STUDY DESIGN:
Intervention Model Description: Enrollment will be initiated with a sentinel cohort of 5 participants randomized to receive DuoChol. The participants in sentinel cohort will be enrolled sequentially one after another after the 2-hour observation period is completed before the next participant is vaccinated. Once 5 participants have received DuoChol, enrollment will be paused until 24-hour safety data is available for all 5 and has been reviewed by the Safety Monitoring Committee (SMC). If no halting criteria defined in the study protocol have been met and the SMC gives approval, enrollment will continue unrestricted.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DuoChol (Experimental): 2 doses of DuoChol capsule administered orally 14 days apart (Day 0 and Day 14).
  Interventions: Biological: DuoChol
- Dukoral® (Active Comparator): 2 doses of Dukoral® administered orally 14 days apart (Day 0 and Day 14). Vaccine suspension is mixed with the buffer (sodium hydrogen carbonate) solution, supplied as effervescent powder.
  Interventions: Biological: Dukoral®

INTERVENTIONS:
Biological: DuoChol — A lyophilized formulation in capsule form (approximately 150mg) contains: - 0.9 mg in 1:1 ratio of formalin inactivated bacteria of two isogenic V. cholerae O1 El Tor strains: serotype Inaba (MS1955) and serotype Ogawa (MS1987) - 0.9 mg of recombinant cholera toxin B subunit (rCTB).
  Arms: DuoChol
Biological: Dukoral® — 3 ml of suspension in a vial contains:
  * 31.25x10^9 bacteria* (approximately) of each of the following V. cholerae O1 strains: Inaba classical biotype (heat inactivated), Inaba El Tor biotype (formalin inactivated), Ogawa classical biotype (heat inactivated), Ogawa classical biotype (formalin inactivated)
  * 1 mg Recombinant cholera toxin B subunit (rCTB)
  5.6 g of effervescent powder (buffer) in a sachet contains Sodium hydrogen carbonate, citric acid, sodium carbonate, saccharin sodium, sodium citrate and raspberry flavor.
  Arms: Dukoral®

SUMMARY:
The goal of this phase I, open-label, randomized, active-controlled Trial is to evaluate the safety and immunogenicity of the DuoChol Oral Cholera Vaccine in 18 to 45 years old healthy participants in Sweden. This first-in-human study is intended to obtain initial data on the DuoChol oral cholera vaccine safety and its effect on immune responses in a cholera non-endemic setting to guide future studies in cholera endemic population. The Investigators will evaluate the safety and immunogenicity after each dose vaccination of DuoChol Oral Cholera Vaccine/Dukoral®.

The participants will be randomly assigned to receive 2 vaccinations at 14-day intervals of DuoChol or Dukoral® in a 2:1 ratio. Participants in the DuoChol arm will receive one capsule of DuoChol on days 0 and 14. Participants in the Dukoral® arm will receive the standard dose as indicated in the Dukoral® package insert. The Investigators will follow-up the participants for 4 weeks after the second vaccination.

The study is funded by Wellcome Trust, grant number : 226726/Z/22/Z.

DETAILED DESCRIPTION:
A total of 60 healthy participants aged 18-45 in Sweden will be recruited and randomly assigned in a 2:1 ratio: 40 participants will receive DuoChol, 20 participants will receive Dukoral®. Each person will receive two doses of DuoChol or Dukoral® orally. There participants will have 6 scheduled study visits, including blood sampling for immunogenicity testing and safety assessment.

Blood samples will be taken at screening, and then during the study, to check immune response and overall health status. Baseline tests include HIV, hepatitis, complete blood counts, and liver function test. Women of childbearing age will undergo pregnancy testing during screening and prior to each vaccination.

All participants will be observed after vaccination for immediate reactions. Serious adverse events will be reported, and followed up till resolution, and participants are instructed to contact the Investigator team if they experience any serious adverse event.

Study Objectives:

* Primary: To evaluate the safety after each dose vaccination of DuoChol Oral Cholera Vaccine.
* Secondary: To compare the immune response of DuoChol with the existing vaccine Dukoral® to assess whether DuoChol can generate a response in the immune system to protect against the disease.

Key Endpoints:

* Monitor for any serious adverse events like hospitalization, death, or significant disability that happen during the study that may or may not be related to the vaccines.
* Track immediate reactions within 1-2 hours after vaccination to detect allergic or other immediate responses.
* Record mild to moderate side effects such as nausea, fever, or diarrhea for up to 14 days after each dose.
* Measure immune response in the blood 14 days after each dose.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female participants aged 18 to 45 years, inclusive, at the time of signing the informed consent.
2. Must have a Swedish (or other nationality) identity card
3. Must be able to understand the information included in the informed consent form and be willing to provide voluntary informed consent to participate in the study
4. Must agree to not take any medication affecting gastric acidity (such as proton pump inhibitor, H2 receptor blocker, or antacid) for 7 days prior to and until 24 hours after each vaccination.
5. Must be able to attend all scheduled study visits and comply with all study procedures.
6. Must be in good general health and without clinically significant medical history, as determined by the study investigator using clinical judgement after review of medical history, physical examination, and laboratory screening tests (hematology, renal function, and liver function tests).
7. Female-Specific Criteria:

   1. Not currently pregnant or breastfeeding and not planning to become pregnant for at least 12 weeks after last vaccination.
   2. Negative urine pregnancy test at the time of vaccination.
   3. Agree to use at least one acceptable an adequate birth control method for at least 4 weeks prior to receipt of vaccine and for at least 12 weeks after receipt of the vaccine. Adequate birth control is defined as follows: Contraceptive medications delivered orally, intramuscularly, vaginally, or implanted underneath the skin, surgical methods (hysterectomy or bilateral tub l ligation), condoms, diaphragms, intrauterine device, or abstinence
8. Male-Specific Criteria:

   1. Be willing to use an adequate birth control method during study participation and 12 weeks after the last vaccination.
   2. For non-vasectomized male participants with female partners of child- bearing potential this includes the use of condoms or abstinence and/or their partner's use of contraceptive medications delivered orally, intramuscularly, vaginally, or implanted underneath the skin, surgical methods (hysterectomy or bilateral tubal ligation), diaphragms, or intrauterine device.

Exclusion Criteria:

1. Any clinically significant symptom of acute illness (e.g., cough, sore throat), febrile illness (tympanic temperature >38°C) within 72 hours prior to the enrollment. A prospective participant should not be included until 72 hours after the condition has completely resolved.
2. Participant with diarrhea, abdominal pain or vomiting in the past 24 hours or with history of diarrhea lasting for more than 2 weeks in the past 6 months.
3. Known history of any immunocompromised condition, including immunodeficiency disease, renal function disorder, malignancy, chronic inflammatory disease, etc.
4. Use of systemic steroids within past 6 months (>10 mg/day prednisone equivalent for period exceeding 2 consecutive weeks), or history of having received chemotherapy, radiation therapy or other immunosuppressive drugs within the past 6 months.
5. Participant who has ever received previous immunization with cholera vaccine, who has received any vaccine within 4 weeks prior to the first dose of study vaccination, or who plans to receive any other vaccine within 4 weeks following last dose of the investigational product.
6. Participant concomitantly enrolled or scheduled to be enrolled in another trial.
7. Participant with previous history of confirmed cholera, salmonella, shigella or ETEC disease.
8. Known history or allergy to vaccine components, or any other allergies deemed by the investigator to increase risk of an adverse event during trial participation.
9. Individuals with a known bleeding disorder, or any condition that may be associated with a prolonged bleeding time resulting in contraindication for blood sample collection.
10. Receipt of blood, blood-derived products, or immunoglobulin products in the past 3 months.
11. Any abnormality or chronic disease which in the opinion of the investigator might be detrimental for the safety of the participant or interfere with the assessment of the study objectives.
12. Any female participant who is lactating*, pregnant, or planning for pregnancy during study period.
13. Individuals who are involved in DuoChol Clinical trial or family/household members of research staff.
14. Any other condition which, in the opinion of the investigator, might interfere with the evaluation of the study objectives (e.g., alcohol or drug abuse, neurologic or psychiatric conditions etc.).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Safety of each investigational product dose at a specified duration | From enrollment to the end of study, approximately 6 weeks for each participant.
  1. Occurrence of any SAEs from the first dose vaccination until 28 days after the second dose vaccination.
  2. Occurrence of immediate adverse events within 2 hours after the first dose of vaccination for the sentinel cohort of participants, and within 1 hour for the rest of the participants
  3. Occurrence of solicited gastrointestinal and systemic adverse events within 7 days after each vaccination
  4. Occurrence of unsolicited adverse events within 14 days after each vaccination
  5. Occurrence of clinically significant changes in safety laboratory parameters after each vaccination

SECONDARY OUTCOMES:
Proportion of participants achieving seroconversion of serum vibriocidal antibody titers against V. cholerae O1 Inaba and V. cholerae O1 Ogawa. | Baseline (prior to first vaccination) to 14 days after the first and second vaccination.
  seroconversion of serum vibriocidal antibody titers defined as at least 4-fold increase
Geometric Mean Titer (GMT) of serum vibriocidal antibody titers against V. cholerae O1 Inaba and V. cholerae O1 Ogawa. | Baseline (prior to first vaccination) to 14 days after the first and second vaccination.
Geometric Mean Fold Rise (GMFR) of serum vibriocidal antibody titers against V. cholerae O1 Inaba and V. cholerae O1 Ogawa. | Baseline (prior to first vaccination) to 14 days after the first and second vaccination.
Proportion of participants achieving seroconversion of serum IgG anti-CTB antibodies. | Baseline (prior to first vaccination) to 14 days after the first and second vaccination.
  seroconversion of serum IgG anti-CTB antibodies defined as at least 2-fold increase
Geometric Mean Titer (GMT) of serum IgG anti-CTB antibodies. | Baseline (prior to first vaccination) to 14 days after the first and second vaccination.
Geometric Mean Fold Rise (GMFR) of serum IgG anti-CTB antibodies. | Baseline (prior to first vaccination) to 14 days after the first and second vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Cowden, MD, Principal Investigator — International Vaccine Institute
Locations (1):
- Studieenheten Akademiskt Specialistcentrum, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No
Restrictions under data protection frameworks (e.g., GDPR) that impose strict requirements on the use, transfer, and sharing of health-related data. The informed consent form does not cover participant agreement for data sharing beyond the purpose or jurisdiction described in the participant's information sheet.